CLINICAL TRIAL: NCT01394939
Title: A Phase 1/2a Dose-escalation Study of JX 594 Administered by Multiple Intravenous (IV) Infusions Alone and in Combination With Irinotecan in Patients With Metastatic, Refractory Colorectal Carcinoma.
Brief Title: Recombinant Vaccinia Virus Administered Intravenously in Patients With Metastatic, Refractory Colorectal Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jennerex Biotherapeutics (Industry)
Collaborators: Transgene (Industry)
Responsible Party: Sponsor
Organization: SillaJen, Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JX594-CRC019
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Carcinoma; CRC
Keywords: Vaccinia; Vaccinia Virus; JX-594; Jennerex; Colorectal Carcinoma; Colorectal cancer; Colon Cancer; Rectal Cancer; oncolytic virus; viral therapy; RAS mutant; Erbitux failure; Oxaliplatin failure; FOLFOX failure; FOLFIRI failure; Irinotecan failure; Pexa-Vec
MeSH Terms: conditions — Colorectal Neoplasms; Vaccinia; Colonic Neoplasms; Rectal Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single Agent_ Cohort 1 (Experimental): JX-594 administered intravenously weekly for 5 weeks followed by up to 3 additional intravenous infusion boosts.
  JX-594: Recombinant Vaccinia Granulocyte-Macrophage Colony-Stimulating Factor (RAC VAC GM-CSF) Cohort 1: JX-594 3 x 10^8 plaque forming unit (pfu), Days 1, 8,15, 22, and 29
  Interventions: Biological: JX-594
- Single Agent_Cohort 2 (Experimental): JX-594 administered intravenously weekly for 5 weeks followed by up to 3 additional intravenous infusion boosts.
  JX-594: RAC VAC GM-CSF Cohort 2: JX-594 1 x 10^9 pfu, Days 1, 8,15, 22, and 29
  Interventions: Biological: JX-594
- Combination_Cohort 3 (Experimental): JX-594 administered intravenously weekly for 5 weeks followed by up to three additional intravenous infusion boosts in combination with Irinotecan administered every 14 days beginning at Day 9.
  JX-594: RAC VAC GM-CSF Irinotecan: 180 mg/m2 IV every 2 weeks. JX-594 3 x 10^8 pfu Day 1,8, 15, 22, 29 + irinotecan 180 mg/m2 biweekly starts on Day 9.
  Interventions: Biological: JX-594; Drug: Irinotecan
- Combination_Cohort 4 (Experimental): JX-594 administered intravenously weekly for 5 weeks followed by up to three additional intravenous infusion boosts in combination with Irinotecan administered every 14 days beginning at Day 9.
  JX-594: RAC VAC GM-CSF JX-594 1 x 10^9 pfu Day1, 8, 15, 22, 29 + irinotecan 180 mg/m2 biweekly starts on Day 9.
  Interventions: Biological: JX-594; Drug: Irinotecan

INTERVENTIONS:
Biological: JX-594 — Recombinant Vaccinia GM-CSF; RAC VAC GM-CSF (JX-594)
Drug: Irinotecan — 180 mg/m2 IV every 2 weeks.
  Arms: Combination_Cohort 3; Combination_Cohort 4

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of JX-594 (Pexa-Vec) administered intravenously either alone or in combination with Irinotecan in colorectal carcinoma patients who are refractory to or intolerant to standard therapy.

DETAILED DESCRIPTION:
This was a Phase 1/2a, open-label, dose-escalation study in patients with advanced colorectal cancer (CRC)

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, advanced metastatic colorectal cancer failed treatment with fluoropyrimidine (fluoruracil or capecitabine) and oxaliplatin based therapies or had contradictions to treatment with these drugs as determined by the investigator
* Failed treatment with irinotecan
* Kras mutant tumor or Kras wild-type having failed cetuximab (Erbitux) or panitumumab (Vectibix) or had contradictions to treatment
* Regorafenib-naïve (have not received regorafenib)
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1 or 2
* Measurable tumor (≥1 cm longest diameter)
* Acceptable health status as determined by the investigator and blood work (Chemistry, Complete Blood Count, Coagulation)

Exclusion Criteria:

* Intolerant to Irinotecan (if assigned to the combination arm: Cohort 3, Cohort 4 or Combination Expansion Arm)
* Treatment with ketoconazole, enzyme-inducing anticonvulsants and St. John's Wort (if assigned to combination arm)
* Significant immunodeficiency due to underlying illness and/or medication
* History of severe exfoliative skin condition requiring systemic therapy within the past 2 years
* Clinically significant and/or rapidly accumulating ascites, pericardial and/or pleural effusions
* Active cardiovascular disease, including but not limited to significant coronary artery disease (e.g., requiring angioplasty or stenting) or congestive heart failure within the preceding 12 months
* Viable Centrual Nervous System (CNS) malignancy associated with clinical symptoms
* Received anti-cancer therapy within 4 weeks prior to first treatment (6 weeks for mitomycin c or nitrosoureas)
* Prior participation in any other research protocol involving an investigational medicinal product within 4 weeks prior to first treatment
* Use of prohibited anti-viral medication, interferon/pegylated interferon (PEG-IFN) or ribavirin that cannot be discontinued within 14 days prior to any JX 594 dose
* Inability to suspend treatment with anti-hypertensive medication for 48 hours prior to and 48 hours after all JX-594 treatments.
* Pregnant or nursing an infant
* Diagnosis of chronic inflammatory bowel disease and/or bowel obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Burke, MD, Study Director — Jennerex Biotherapeutics; Derek Jonker, MD, Principal Investigator — Ottawa Hospital and Research Institute
Locations (11):
- United States (6):
  - Mayo Clinic, Scottsdale, Arizona
  - UCSD Moores Cancer Center, La Jolla, California
  - Billings Clinic Cancer Center, Billings, Montana
  - University of North Carolina, Chapel Hill, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - The Ohio State University, Columbus, Ohio
- Canada (2):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Ottawa Hospital and Research Institute (OHRI), Ottawa, Ontario
- France (3):
  - Hôpital Saint Antoine, Paris
  - Hôpital Hautepierre, Strasbourg
  - Institut Claudius Regaud, Toulouse

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 patients out of 52 enrolled experienced no study related Adverse Event (AE) and was not included in the started population.
Groups:
- Single Agent_ Cohort 1: JX-594 administered intravenously weekly for 5 weeks followed by up to 3 additional intravenous infusion boosts.
  Cohort 1: JX-594 3 x 10^8 pfu, Days 1, 8,15, 22, and 29
- Single Agent_Cohort 2: JX-594 administered intravenously weekly for 5 weeks followed by up to 3 additional intravenous infusion boosts.
  Cohort 2: JX-594 1 x 10^9 pfu, Days 1, 8,15, 22, and 29
- Combination_Cohort 3: JX-594 administered intravenously weekly for 5 weeks followed by up to three additional intravenous infusion boosts in combination with Irinotecan administered every 14 days beginning at Day 9.
  Irinotecan: 180 mg/m2 IV every 2 weeks.
  JX-594 3 x 10^8 pfu Day 1,8, 15, 22, 29 + irinotecan 180 mg/m2 biweekly starts on Day 9.
- Combination_Cohort 4: JX-594 administered intravenously weekly for 5 weeks followed by up to three additional intravenous infusion boosts in combination with Irinotecan administered every 14 days beginning at Day 9.
  JX-594 1 x 10^9 pfu Day1, 8, 15, 22, 29 + irinotecan 180 mg/m2 biweekly starts on Day 9.
Period: Overall Study
Arm/Group | Single Agent_ Cohort 1 | Single Agent_Cohort 2 | Combination_Cohort 3 | Combination_Cohort 4
Started | 4 | 25 | 4 | 17
Completed | 3 | 15 | 4 | 10
Not Completed | 1 | 10 | 0 | 7
Not completed — Adverse Event | 1 | 3 | 0 | 2
Not completed — Death | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 2
Not completed — Others | 0 | 2 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Single Agent_ Cohort 1: JX-594 administered intravenously weekly for 5 weeks followed by up to 3 additional intravenous infusion boosts.
  JX-594 3 x 10^8 pfu, Days 1, 8,15, 22, and 29
- Single Agent_Cohort 2: JX-594 administered intravenously weekly for 5 weeks followed by up to 3 additional intravenous infusion boosts.
  JX-594 1 x 10^9 pfu, Days 1, 8,15, 22, and 29
- Combination_Cohort 3: JX-594 administered intravenously weekly for 5 weeks followed by up to three additional intravenous infusion boosts in combination with Irinotecan administered every 14 days beginning at Day 9.
  JX-594 3 x 10^8 pfu Day 1,8, 15, 22, 29 + irinotecan 180 mg/m2 biweekly starts on Day 9.
- Total: Total of all reporting groups
Arm/Group | Single Agent_ Cohort 1 | Single Agent_Cohort 2 | Combination_Cohort 3 | Combination_Cohort 4 | Total
Number analyzed (Participants) | 4 | 25 | 4 | 17 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 15 | 3 | 10 | 31
  >=65 years | 1 | 10 | 1 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (8.06) | 58.3 (11.84) | 58.8 (13.74) | 58.6 (10.42) | 58.9 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 13 | 1 | 6 | 20
  Male | 4 | 12 | 3 | 11 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 25 | 4 | 15 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 3 | 3
  White | 4 | 25 | 4 | 11 | 44
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Determine Radiographic Response Rate of Patients Enrolled in the Phase 2a Portion of the Study
Description: Percentage of participants who showed overall response during their participation in the study. Per Modified Response Evaluation Criteria In Solid Tumors Criteria (mRECIST) and assessed by tri-phasic contrast enhanced CT: Complete Response (CR), Disappearance of intratumoral enhancing area; Partial Response (PR), >=30% decrease in the sum of the diameters of enhancing area; Overall Response (OR) = CR + PR.
Time Frame: Scans Every 8 weeks until radiographic progression was confirmed by the site.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Agent_ Cohort 1 | Single Agent_Cohort 2 | Combination_Cohort 3 | Combination_Cohort 4
Number analyzed (Participants) | 4 | 25 | 4 | 17
Participants | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Single Agent_ Cohort 1: JX-594 administered intravenously weekly for 5 weeks followed by up to 3 additional intravenous infusion boosts.
  JX-594: Recombinant Vaccinia GM-CSF; RAC VAC GM-CSF (JX-594)
  Cohort 1: Pexa-Vec 3 x 108 pfu, Days 1, 8,15, 22, and 29
- Single Agent_Cohort 2: JX-594 administered intravenously weekly for 5 weeks followed by up to 3 additional intravenous infusion boosts.
  JX-594: Recombinant Vaccinia GM-CSF; RAC VAC GM-CSF (JX-594)
  Cohort 2: Pexa-Vec 3 x 109 pfu, Days 1, 8,15, 22, and 29
- Combination_Cohort 3: JX-594 administered intravenously weekly for 5 weeks followed by up to three additional intravenous infusion boosts in combination with Irinotecan administered every 14 days beginning at Day 9.
  JX-594: Recombinant Vaccinia GM-CSF; RAC VAC GM-CSF (JX-594)
  Irinotecan: 180 mg/m2 IV every 2 weeks.
  Cohort 3: Pexa-Vec 3 x 108 pfu Day 1,8, 15, 22, 29 + irinotecan 180 mg/m2 biweekly starts on Day 9.
- Combination_Cohort 4: JX-594 administered intravenously weekly for 5 weeks followed by up to three additional intravenous infusion boosts in combination with Irinotecan administered every 14 days beginning at Day 9.
  JX-594: Recombinant Vaccinia GM-CSF; RAC VAC GM-CSF (JX-594)
  Cohort 4: Pexa-Vec 1 x 109 pfu Day1, 8, 15, 22, 29 + irinotecan 180 mg/m2 biweekly starts on Day 9.
Arm/Group | Single Agent_ Cohort 1 | Single Agent_Cohort 2 | Combination_Cohort 3 | Combination_Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/4 | 2/25 | 0/4 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/4 | 10/25 | 1/4 | 8/17
Other Adverse Events (participants affected / at risk) | 4/4 | 25/25 | 4/4 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent_ Cohort 1 (N=4) | Single Agent_Cohort 2 (N=25) | Combination_Cohort 3 (N=4) | Combination_Cohort 4 (N=17)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 2 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pelvic infection (Infections and infestations) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 1 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent_ Cohort 1 (N=4) | Single Agent_Cohort 2 (N=25) | Combination_Cohort 3 (N=4) | Combination_Cohort 4 (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 6 | 2 | 6
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 6 | 3 | 7
Ventricular hypokinesia (Cardiac disorders) | 1 | 0 | 0 | 0
Eyepain (Eye disorders) | 0 | 1 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 4 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 7 | 2 | 5
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 3 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 2 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 13 | 4 | 14
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 12 | 4 | 10
Asthenia (General disorders) | 0 | 2 | 0 | 0
Catheter site pruritus (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 4 | 19 | 4 | 15
Device occlusion (General disorders) | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 2 | 7 | 4 | 12
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 2 | 1 | 0
Injection site pain (General disorders) | 1 | 1 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 2 | 0
Mass (General disorders) | 0 | 1 | 0 | 0
Medical device complication (General disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 3
Oedema peripheral (General disorders) | 1 | 7 | 3 | 4
Pain (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 4 | 23 | 4 | 17
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 2 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 3
Pelvic infection (Infections and infestations) | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 3 | 11 | 1 | 6
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 2
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Splinter (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 3 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 3 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 4 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 8 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 3 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2
Red blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 3 | 0 | 2
Weight increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4 | 4 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 2
Dysaesthesia (Nervous system disorders) | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Extensor plantar response (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 12 | 3 | 7
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 3
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Encopresis (Psychiatric disorders) | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 1 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 6
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Capillaritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 5 | 2 | 7
Hypotension (Vascular disorders) | 2 | 16 | 3 | 11
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No